CLINICAL TRIAL: NCT06159361
Title: The Effect of a Targeted Exercise Program on Balance and Postural Responses in Patients With Multiple Sclerosis (MS)
Brief Title: Balance Targeted Exercises for Individuals With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, James Moore, Associate professor of clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231151
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance targeted exercises group (Experimental): participants in this group will receive the balance targeted exercises for up to 6 weeks
  Interventions: Behavioral: Balance targeted exercises

INTERVENTIONS:
Behavioral: Balance targeted exercises — 6-week exercise program, 3 sessions per week (2 sessions in person, 1 session of home exercises. Participants will receive a booklet with information about the home exercises and will receive a text message reminder), each session will last 60 minutes.

SUMMARY:
The purpose of this study is to examine the effects of a postural adjustment, targeted training program on balance ability and postural responses anticipatory postural adjustments (APA) and compensatory postural adjustments (CPA) in individuals with MS

DETAILED DESCRIPTION:
All participants participated in individual training program aimed at improving balance ability and postural adjustments. The training program and individual activities were based on previously published programs and motor learning principles, and consists of 18, 1-hour training sessions over six weeks (3 sessions/week). Training occurred in person 2 days a week (in person training) and at home (home exercise program) 1 day a week, for a total of 3 sessions per week. The duration of training sessions were 60 minutes per session for a total of 1,140 minutes of training. The exercise room temperature was centrally regulated (23.3 degrees C).

ELIGIBILITY:
Inclusion Criteria:

1. Must be18 to 70 years of age.
2. Medical diagnosis of MS confirmed by a neurologist.
3. Ability to stand independently without any aid for at least 3 minutes.
4. A Patients determined disease steps (PDDS) score of 5 or lower.
5. Normal or corrected-to-normal vision.
6. English or Spanish speaking.

Exclusion Criteria:

1. MS-related exacerbation or medication change in the past two months.
2. Presence of concurrent neurological or orthopedic disorders.
3. Unable to perform the experimental tasks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in balance ability as measured by the BESTest | Baseline, 6 weeks (post intervention)
  The Balance Evaluation Systems Test (BESTest) will be used to measure balance ability. Items are scored from 0 (severe impairment) to 3 (no impairment), with a total score of 108. A higher score suggests better balance ability.
Change in reaction time | Baseline, 6 weeks (post intervention)
  Measure in seconds
Change in movement velocity | Baseline, 6 weeks (post intervention)
  Measure in degree per second
Change in endpoint excursion percentage | Baseline, 6 weeks (post intervention)
  measure of endpoint excursion in a percentage out of a100
Change in directional control percentage | Baseline, 6 weeks (post intervention)
  measure of directional control in a percentage out of a100
Change in maximum excursion percentage | Baseline, 6 weeks (post intervention)
  measure of maximum excursion in a percentage out of a100
Change in muscle responses latency as measured by MCT | Baseline, 6 weeks (post intervention)
  The Motor Control test (MCT) measures the subject's ability to generate a motor response latency to a sudden surface translation in a forward and backward direction at three different magnitudes (small, medium, and large).
  Latency: The time-lapse between the perturbation onset and the subject response for each limb. The latency is reported in milliseconds.
Change in postural muscles responses latency as measured by Electromyography (EMG) | Baseline, 6 weeks (post intervention)
  Postural muscles responses onset latency in seconds
Change in APA as measured by microvolts | Baseline, 6 weeks (post intervention)
  Postural muscles APA measured in microvolts
Change in CPA as measured by microvolts | Baseline, 6 weeks (post intervention)
  Postural muscles CPA in microvolts

SECONDARY OUTCOMES:
Change in balance confidence as measured by ABC | Baseline, 6 weeks (post intervention)
  The Activities Specific Balance Confidence (ABC) scale is a self-report questionnaire of a subject's perceived level of balance confidence. It measures the subject's confidence in performing various ambulatory activities without falling. There are 16 items scored using a scale(0-100) with higher scores indicating more confidence in performing the tasks. A total score is reported by dividing the total ABC score by 16.
Change in quality of life as measured by the MSQoL-54 | Baseline, 6 weeks (post intervention)
  Multiple Sclerosis Quality of Life - 54 (MSQoL-54) is a self-report questionnaire measuring subject perceived of quality of life. In total, it contains 54 items with a total score ranging from 0-100, with higher scores indicating a better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: James Moore, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No